CLINICAL TRIAL: NCT07393789
Title: A Multicomponent Physical Activity Intervention Effect on Weekly Steps and Physical Fitness in Preadolescents: A Pretest-Posttest Study and Randomized Control Trial
Brief Title: A Multicomponent Physical Activity Intervention Effect on Weekly Steps and Physical Fitness in Preadolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Vladimir Milošević, Assistant professor, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COMPASS-2022
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Multicomponent 16-week Program Comprised of a Goal Setting, Wearable Activity Tracker Feedback, Physical Exercising, and Motivating Students to be Active
Keywords: Pretest-Posttest Study; Randomized Control Trial; physical activity intervention, children, preadolescents, physical fitness, body mass index, school-based intervention

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either an intervention group or a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Intervention Group (Experimental): Participants receive a 16-week structured multicomponent physical activity program.
  Interventions: Behavioral: Multicomponent Physical Activity Program
- Control Group (No Intervention): Participants continue their usual daily activities without additional intervention.

INTERVENTIONS:
Behavioral: Multicomponent Physical Activity Program — Structured physical activity sessions and motivational procedures designed to improve muscular strength, cardiorespiratory fitness, speed, and coordination.
  Arms: Physical Activity Intervention Group

SUMMARY:
This study examines the effects of a 16-week structured physical activity program on physical fitness, steps number, and body mass index in children aged 8 to 10 years.

Participants were randomly assigned to either an intervention group that participated in the physical activity program or a control group that continued with their usual daily activities without additional intervention.

Physical fitness outcomes include standing broad jump, handgrip strength, and 20-meter shuttle run performance. Body mass index is calculated from measured height and body mass.

The goal of the study is to determine whether participation in a multicomponent physical activity intervention leads to greater improvements in physical fitness, steps number, and body composition compared with no additional intervention.

DETAILED DESCRIPTION:
This randomized controlled trial investigated the effects of a multicomponent physical activity intervention on physical fitness, steps number, and body mass index in preadolescent children.

Children aged 8 to 10 years were recruited from a primary school setting and randomly allocated to either an intervention group or a control group. The intervention group participated in a structured physical activity program and motivational strategies lasting 16 weeks, while the control group continued their regular daily routines and school activities without additional intervention activities provided by the study.

The physical activity program consisted of planned sessions designed to develop muscular strength, cardiorespiratory endurance, speed, and coordination through age-appropriate exercises and games.

Assessments were conducted before and after the intervention period. Physical fitness was evaluated using the standing broad jump (lower-body muscular power), handgrip strength (upper-body muscular strength), and the 20-meter shuttle run test (cardiorespiratory fitness). Body mass index was calculated using measured body mass and height.

The primary objective of the study was to determine whether children participating in the intervention demonstrate greater improvements in physical fitness and body mass index compared with children in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 8 to 10 years.
* Enrollment in regular primary school.
* Written informed consent obtained from parent or legal guardian.
* Ability to participate in physical education and physical activity.

Exclusion Criteria:

* Medical conditions or physical disabilities that limit participation in physical activity.
* Acute illness or injury at the time of testing.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 178 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Handgrip Strength | Baseline and 16 weeks
  Handgrip Strength in kg
Standing Broad Jump Distance | Baseline and 16 weeks
  Assessment of lower-body muscular power measured in centimeters
20-Meter Shuttle Run Performance | Baseline and 16 weeks
  20-Meter Shuttle Run result in seconds

SECONDARY OUTCOMES:
Body Mass Index (BMI) | Baseline and 16 weeks
  BMI is calculated by dividing weight in kilograms by height in meters squared.

CONTACTS AND LOCATIONS:
Locations (2):
- Zakladni skola Travnik, Přerov, Czechia
- University of Belgrade - Faculty of Sport and Physical Education, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No